CLINICAL TRIAL: NCT05831254
Title: Comparison of the Effects of European Health Literacy Based Education and E-Pulse Education on the Level of Health Literacy in Adults Aged 45-64: a Randomized Controlled Study with Active Control Group
Brief Title: The Effect of Health Literacy Education in Adults (HELP-e-Pulse)
Acronym: HELP-e-Pulse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Sebahat Gozum, Prof.Dr.Sebahat Gozum, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 003
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-04

CONDITIONS: Health Literacy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HEalth Literacy, e-Pulse (HELP) (Experimental)
  Interventions: Other: Health education:Interactive group training
- e-Pulse (Active Comparator)
  Interventions: Other: Health education: Individually training

INTERVENTIONS:
Other: Health education:Interactive group training — 1. To introduce e-pulse software, which is a personal health record system, to show its use, to provide training materials such as video-brochures about e-pulse. This program will be done as interactive group training
  2. Six modular interactive group training, each of which includes the steps of the European Health Literacy Scale of 90 minutes.
  Arms: HEalth Literacy, e-Pulse (HELP)
Other: Health education: Individually training — To introduce e-pulse software, which is a personal health record system, to provide training materials such as video-brochures about e-pulse. This education will be done individually.
  Arms: e-Pulse

SUMMARY:
The world's elderly population is increasing. It is possible to prepare for the old age period by starting to develop the level of Health Literacy (HL) in the 45-64 age group. In this context, this study is planned to be conducted as a randomized controlled study with an active control group in order to compare the effect of European Health Literacy-based education and e-Pulse education (HELP) on the level of health literacy in adults aged 45-64 with insufficient-limited health literacy. The study was planned to include a total of 140 participants from the intervention group (HELP) (n:70) and the active control group (e-Pulse) (n:70). Interactive group training consisting of six modules and 90 minutes each will be given to the HELP group. Individual e-Pulse instruction will be given to the active control group. European Health Literacy Scale scores will be considered as the primary outcome of the research. Scores from the eHealth Literacy Scale will be considered as the secondary outcome of the research.

ELIGIBILITY:
Inclusion Criteria:

* Being aged 45-64 and above and being literate,
* Having a score of 33 or less on the European Health Literacy Scale (insufficient, limited and problematic health literacy)
* Being able to use a smart phone, tablet or computer,
* Having agreed to voluntarily participate in the study.

Exclusion Criteria:

• Those who do not speak Turkish

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
European Health Literacy Scale | Baseline-Second month
  This scale is a self-report measure used to evaluate the health literacy level for individuals over 15 years old. It includes three topics (treatment, prevention from diseases and improving health) and 47 items. Each item has four possible answers: 1 = Very difficult, 2 = Difficult, 3 = Easy and 4 = Very easy. A 'Don't know' answer is coded as 5. Health literacy level is evaluated in four categories according to the score obtained: (0-25) points: insufficient health literacy; (>25-33) : problematic - limited health literacy; (>33-42) : adequate health literacy; (>42-50) : indicates excellent health literacy.

SECONDARY OUTCOMES:
eHealth Literacy Scale | Baseline-Second month
  The eHEALS is an 8-item measure of eHealth literacy developed to measure consumers' combined knowledge, comfort, and perceived skills at finding, evaluating, and applying electronic health information to health problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Soğuksu Yaşlı Evi, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gozum S, Asi E, Siklaroglu M, Sahin S, Oncel S, Imamoglu D, Kanli S. The Effect of European Health Literacy-Based e-Pulse Education and e-Pulse Instructional Materials on Health Literacy Levels in Adults Aged 45-64: A Randomized Controlled Trial. Res Nurs Health. 2025 Jun;48(3):324-336. doi: 10.1002/nur.22450. Epub 2025 Jan 30. PMID 39887466